CLINICAL TRIAL: NCT03243708
Title: Title: EHR Embedded Risk Calculator vs. Standard VTE Prophylaxis for Medical Patients
Brief Title: Title: Randomized Trial of an EHR Embedded Risk Calculator vs. Standard VTE Prophylaxis for Medical Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Michael Rothberg, Staff Physician, The Cleveland Clinic
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 17-396
Record Dates: First submitted 2017-07-10; First posted 2017-08-09 (Actual); Last update posted 2019-05-24 (Actual); Status verified 2019-05

CONDITIONS: Venous Thromboembolism
Keywords: Venous Thromboembolism Risk Calculator
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Intervention Model Description: Step-Wedge Randomized controlled trial (RCT)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Control: Standard order set without risk calculator (usual care)
- Risk calculator (Active Comparator): Intervention: VTE risk calculator embedded in the smart order set incorporated into the EHR and activated for all medical patients
  Interventions: Behavioral: Risk calculator

INTERVENTIONS:
Behavioral: Risk calculator — Venous thromboembolism (VTE) risk calculator embedded in the admission order set with personalized recommendation for prophylaxis
  Arms: Risk calculator

SUMMARY:
Venous thromboembolism (VTE) is a serious source of hospital morbidity and mortality. Chemoprophylaxis with heparin has been shown to reduce the occurrence of VTE, but it increases the risk of bleeding and it is uncomfortable to receive. For that reason, VTE prophylaxis should be reserved for patients at moderate to high risk of VTE and low risk of bleeding. However, identifying patients at low risk for VTE can be difficult, because most patients have at least one risk factor for VTE and there are no validated risk prediction tools for use in US hospitals. Instead, many hospitals have opted for a one-size-fits-all approach with near-universal prophylaxis, putting many patients at unnecessary risk of bleeding. However, to provide care that is truly patient-centered, US physicians face several challenges. First, there is no accepted risk calculator that they can use to estimate an individual patient's risk. Second, risk calculators are not readily available at the point of care. As a result, prophylaxis rates have remained stubbornly low in some institutions, while in others the rate of prophylaxis is high, but the rate of inappropriate prophylaxis is also high. This study uses a risk prediction tool developed at the Cleveland Clinic to assess an individual patient's risk of VTE. The tool is incorporated into the electronic health record in the form of a smart order set. In this randomized trial, we will assess the effects of the order set on physician behavior and patient outcomes . Examining the effectiveness of an electronic decision aid embedded in an EHR in routine clinical practice will test whether a smart order set can improve patient care by incorporating patient-specific factors into a complex decision process.

DETAILED DESCRIPTION:
Specific Aim:

Assess the effects of a VTE risk calculator embedded in the admission order set vs. usual care on physician behavior and patient outcomes in a randomized trial

Research Strategy:

Utilizing a Step-Wedge design, this randomized controlled trial (RCT) will be conducted at 10 Cleveland Clinic hospitals in efforts to assess the effects of a VTE (venous thromboembolism) risk calculator embedded in the admission order set vs. usual care on physician behavior and patient outcomes. Hospitals will be randomized to display the risk calculator to physicians admitting patients or to the usual order set that contains only a description of VTE risk factors. The risk calculator will produce a predicted risk of VTE together with a recommendation regarding the use of prophylaxis for an individual patient. Physicians will be free to ignore the calculator or override its results if they so choose.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients (age ≥18 years) admitted to a medical service, including intensive care units, between September 1, 2017 and August 31, 2018 will be eligible.

Exclusion Criteria:

* patients not eligible to receive VTE prophylaxis because they are already receiving anticoagulation for another purpose (e.g. warfarin for atrial fibrillation or LMWH for DVT or PE present on admission),
* patients admitted with a terminal condition who are receiving comfort care only
* Surgical patients who are admitted to the medical service temporarily (e.g. hip fracture)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90537 (Actual)
Dates: Start 2017-12-04 (Actual); Primary Completion 2019-04-14 (Actual); Study Completion 2019-04-14 (Actual)

PRIMARY OUTCOMES:
Appropriate VTE prophylaxis | within 48 hours of index hospitalization admission
  Proportion of patients at high risk of VTE who receive prophylaxis and the proportion of patients at low risk who do not receive prophylaxis

SECONDARY OUTCOMES:
Total patients receiving prophylaxis | 14 days
  All patients who received any chemoprophylaxis during hospitalization, regardless of risk status.
Rate of VTE among high risk patients | 14 days
  Symptomatic VTE events not present on admission occurring among patients at high risk for VTE according to the risk calculator.
Rate of VTE among high risk patients | 45 days
  Symptomatic VTE events not present on admission occurring among patients at high risk for VTE according to the risk calculator.
Rate of major bleeding among high risk patients | 14 days
  Major bleeding events among patients with risk factors for bleeding.
Average cost of prophylaxis | 14 days
  Total cost of prophylaxis received during hospitalization
Average cost of hospitalization | Up to 30 days
  Cost of hospitalization as determined by the hospital cost accounting system
Average length of stay | Up to 30 days
  Total days in hospital

CONTACTS AND LOCATIONS:
Overall Officials: Michael Rothberg, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Health System, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lederle FA, Zylla D, MacDonald R, Wilt TJ. Venous thromboembolism prophylaxis in hospitalized medical patients and those with stroke: a background review for an American College of Physicians Clinical Practice Guideline. Ann Intern Med. 2011 Nov 1;155(9):602-15. doi: 10.7326/0003-4819-155-9-201111010-00008. PMID 22041949
- [Background] Kakkar AK, Cimminiello C, Goldhaber SZ, Parakh R, Wang C, Bergmann JF; LIFENOX Investigators. Low-molecular-weight heparin and mortality in acutely ill medical patients. N Engl J Med. 2011 Dec 29;365(26):2463-72. doi: 10.1056/NEJMoa1111288. PMID 22204723
- [Background] Rothberg MB, Lahti M, Pekow PS, Lindenauer PK. Venous thromboembolism prophylaxis among medical patients at US hospitals. J Gen Intern Med. 2010 Jun;25(6):489-94. doi: 10.1007/s11606-010-1296-y. Epub 2010 Mar 30. PMID 20352366
- [Background] Cohen AT, Tapson VF, Bergmann JF, Goldhaber SZ, Kakkar AK, Deslandes B, Huang W, Zayaruzny M, Emery L, Anderson FA Jr; ENDORSE Investigators. Venous thromboembolism risk and prophylaxis in the acute hospital care setting (ENDORSE study): a multinational cross-sectional study. Lancet. 2008 Feb 2;371(9610):387-94. doi: 10.1016/S0140-6736(08)60202-0. PMID 18242412
- [Background] Khanna R, Vittinghoff E, Maselli J, Auerbach A. Unintended consequences of a standard admission order set on venous thromboembolism prophylaxis and patient outcomes. J Gen Intern Med. 2012 Mar;27(3):318-24. doi: 10.1007/s11606-011-1871-x. Epub 2011 Sep 24. PMID 21948203
- [Background] Qaseem A, Chou R, Humphrey LL, Starkey M, Shekelle P; Clinical Guidelines Committee of the American College of Physicians. Venous thromboembolism prophylaxis in hospitalized patients: a clinical practice guideline from the American College of Physicians. Ann Intern Med. 2011 Nov 1;155(9):625-32. doi: 10.7326/0003-4819-155-9-201111010-00011. PMID 22041951
- [Background] Barbar S, Noventa F, Rossetto V, Ferrari A, Brandolin B, Perlati M, De Bon E, Tormene D, Pagnan A, Prandoni P. A risk assessment model for the identification of hospitalized medical patients at risk for venous thromboembolism: the Padua Prediction Score. J Thromb Haemost. 2010 Nov;8(11):2450-7. doi: 10.1111/j.1538-7836.2010.04044.x. PMID 20738765
- [Background] Kucher N, Koo S, Quiroz R, Cooper JM, Paterno MD, Soukonnikov B, Goldhaber SZ. Electronic alerts to prevent venous thromboembolism among hospitalized patients. N Engl J Med. 2005 Mar 10;352(10):969-77. doi: 10.1056/NEJMoa041533. PMID 15758007
- [Background] Dunn AS, Brenner A, Halm EA. The magnitude of an iatrogenic disorder: a systematic review of the incidence of venous thromboembolism for general medical inpatients. Thromb Haemost. 2006 May;95(5):758-62. PMID 16676063
- [Background] Bhalla R, Berger MA, Reissman SH, Yongue BG, Adelman JS, Jacobs LG, Billett H, Sinnett MJ, Kalkut G. Improving hospital venous thromboembolism prophylaxis with electronic decision support. J Hosp Med. 2013 Mar;8(3):115-20. doi: 10.1002/jhm.1993. Epub 2012 Nov 26. PMID 23184857
- [Background] Zeidan AM, Streiff MB, Lau BD, Ahmed SR, Kraus PS, Hobson DB, Carolan H, Lambrianidi C, Horn PB, Shermock KM, Tinoco G, Siddiqui S, Haut ER. Impact of a venous thromboembolism prophylaxis "smart order set": Improved compliance, fewer events. Am J Hematol. 2013 Jul;88(7):545-9. doi: 10.1002/ajh.23450. Epub 2013 Jun 12. PMID 23553743
- [Background] Baio G, Copas A, Ambler G, Hargreaves J, Beard E, Omar RZ. Sample size calculation for a stepped wedge trial. Trials. 2015 Aug 17;16:354. doi: 10.1186/s13063-015-0840-9. PMID 26282553
- [Background] Shekelle PG, Wachter RM, Pronovost PJ, Schoelles K, McDonald KM, Dy SM, Shojania K, Reston J, Berger Z, Johnsen B, Larkin JW, Lucas S, Martinez K, Motala A, Newberry SJ, Noble M, Pfoh E, Ranji SR, Rennke S, Schmidt E, Shanman R, Sullivan N, Sun F, Tipton K, Treadwell JR, Tsou A, Vaiana ME, Weaver SJ, Wilson R, Winters BD. Making health care safer II: an updated critical analysis of the evidence for patient safety practices. Evid Rep Technol Assess (Full Rep). 2013 Mar;(211):1-945. PMID 24423049
- [Derived] Rothberg MB, Hamilton AC, Hu B, Sheehan M, Fox J, Milinovich A, Lisheba O, Goto T, Speaker SL, Pappas MA. Impact of Embedding a Venous Thromboembolism Risk Assessment Model in the Electronic Health Record Versus Usual Care: A Cluster-Randomized Trial. Circ Cardiovasc Qual Outcomes. 2025 Aug;18(8):e010359. doi: 10.1161/CIRCOUTCOMES.123.010359. Epub 2024 Feb 6. PMID 38318703